CLINICAL TRIAL: NCT03170011
Title: The Effects of the Biodex Sit2Stand Trainer on Function for Individuals With Cardiac Disease
Brief Title: Biodex Sit2Stand for Individuals With Cardiac Disease
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to enroll any participants.
Sponsor: St. Ambrose University (Other)
Responsible Party: Principal Investigator, Michael Puthoff, Professor, St. Ambrose University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2017-05-14; First posted 2017-05-30 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Coronary Artery Disease; Frail Elderly Syndrome; Heart Failure
Keywords: Cardiac rehabilitation; Sit to Stand; Function
MeSH Terms: conditions — Coronary Artery Disease; Heart Failure

STUDY DESIGN:
Intervention Model Description: This cohort design study will examine the effects of a six week training program using the Biodex Sit2Stand Trainer.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): The training protocol will be include 12 sessions completed over six weeks following a periodization training format. Each session will last approximately 40 minutes. At first, training will focus on high volume, low intensity, self-selected velocity with a progression to high intensity, low volume, self-selected velocity ending with a focus on power training (moderate intensity, moderate volume, high velocity movement) over the six weeks of training.
  Interventions: Behavioral: Exercise using the Biodex Sit2Stand Trainer

INTERVENTIONS:
Behavioral: Exercise using the Biodex Sit2Stand Trainer — Week 1-2 - Focused on lower intensity, higher volume, comfortable/self-selected velocity Week 3-4 - Focus on higher intensity, lower volume, comfortable/self-selected velocity Week 5 - Focus on moderate intensity, moderate volume, transitioning to higher velocity Week 6 - Focus on moderate intensity, moderate volume, high velocity
  Other Names: Biodex Sit2Stand Trainer

SUMMARY:
Patients with cardiac disease have been shown to have deficits in activities such as standing up from a chair. The Biodex Sit2Stand Trainer is a new device meant to improve sit to stand performance by providing a lifting force through the seat to help the individual stand. The amount of lift can be graded to help improve leg strength, endurance, and function over time. The device has the potential to be a form of training for those in cardiac rehabilitation who have limitations in standing from a chair.

DETAILED DESCRIPTION:
Patients who are diagnosed with cardiovascular disease and enter cardiac rehabilitation present with limitations in activity and restrictions in their abilities to participate in society. Even after a standard course of cardiac rehabilitation, some individuals will still present with deficits. One area this is seen is the ability to stand up from a chair. A new device, the Biodex Sit2Stand Trainer, has been designed to help improve the standing movement in those with lower extremity weakness. The trainer provides a graded lift or push through the seat to help the participant reach a standing posture. This study will whether a six week training program using the trainer will lead to improvements in strength, function and quality of life for those individuals who have recently completed a cardiac rehabilitation program. This study is a pilot study to help determine the ideal dosage of training and identify any limitations in using the device with this population. Based on the results of this pilot work, a larger intervention study will be conducted to examine the effectiveness of the trainer in a cardiac rehabilitation program.

ELIGIBILITY:
Inclusion Criteria:

Individuals nearing the end of their cardiac rehabilitation program will be asked to participate. Inclusion criteria include the following:

* Completion of a cardiac rehabilitation
* Ability to walk 50 feet independently with or without an assistive device
* Inability to stand from a standard chair five times without the use of their arms or unable to complete five sit to stands in less than 15 seconds.
* No major cardiac arrhythmias during cardiac rehabilitation sessions.
* Ability to attend 14 sessions over a 7-8 week period

Exclusion Criteria:

* Not meeting inclusion criteria

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-06-01 (Estimated); Primary Completion 2017-09-15 (Estimated); Study Completion 2017-09-15 (Estimated)

PRIMARY OUTCOMES:
Change in Short Physical Performance Battery | Week 0 and Week 7
  Lower extremity functional assessment tool which include gait speed, sit to stand ability and static balance

SECONDARY OUTCOMES:
Change in Isometric knee extension strength | Week 0 and Week 7
  Measured in 90 degrees of flexion with hand held dynamometer
Change in 10 meter gait speed | Week 0 and Week 7
  Self selected walking speed over 10 meters
Change in Six Minute Walk Test | Week 0 and Week 7
  Total distance ambulated during a 6 minute time period.
Change in HeartQoL | Week 0 and Week 7
  Quality of Life assessment tool
Change in MacNew | Week 0 and Week 7
  Quality of life assessment tool

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jensen KH, Baekgaard N, Gaardsting O, Jelnes R, Tonnesen KH. [The social consequences of intermittent claudication]. Ugeskr Laeger. 1986 Oct 13;148(42):2715-7. No abstract available. Danish. PMID 3787784
- [Result] Stevenson TG, Riggin K, Nagelkirk PR, Hargens TA, Strath SJ, Kaminsky LA. Physical activity habits of cardiac patients participating in an early outpatient rehabilitation program. J Cardiopulm Rehabil Prev. 2009 Sep-Oct;29(5):299-303. doi: 10.1097/HCR.0b013e3181b4ca61. PMID 19935142
- [Result] Zullo MD, Dolansky MA, Jackson LW. Cardiac rehabilitation, health behaviors, and body mass index post-myocardial infarction. J Cardiopulm Rehabil Prev. 2010 Jan-Feb;30(1):28-34. doi: 10.1097/HCR.0b013e3181c8594b. PMID 20068420
- [Result] Goel K, Shen J, Wolter AD, Beck KM, Leth SE, Thomas RJ, Squires RW, Perez-Terzic CM. Prevalence of musculoskeletal and balance disorders in patients enrolled in phase II cardiac rehabilitation. J Cardiopulm Rehabil Prev. 2010 Jul-Aug;30(4):235-9. doi: 10.1097/HCR.0b013e3181e17387. PMID 20551829
- [Result] Ades PA, Maloney A, Savage P, Carhart RL Jr. Determinants of physical functioning in coronary patients: response to cardiac rehabilitation. Arch Intern Med. 1999 Oct 25;159(19):2357-60. doi: 10.1001/archinte.159.19.2357. PMID 10547176
- [Result] Puthoff ML, Youngs B. Cardiac Rehabilitation Leads to Improvements in Activity Limitations. J Cardiopulm Rehabil Prev. 2017 Nov;37(6):424-427. doi: 10.1097/HCR.0000000000000220. PMID 28033164